CLINICAL TRIAL: NCT04310228
Title: Favipiravir Combined With Tocilizumab in the Treatment of Corona Virus Disease 2019-A Multicenter, Randomized and Controlled Clinical Trial Study
Brief Title: Favipiravir Combined With Tocilizumab in the Treatment of Corona Virus Disease 2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Principal Investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020YFC0844100
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Novel coronavirus pneumonia; Favipiravir; Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; favipiravir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Favipiravir Combined With Tocilizumab group (Experimental): Favipiravir: On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 7 days.
  Tocilizumab:The first dose is 4 ~ 8mg/kg and the recommended dose is 400mg. For fever patients, an additional application (the same dose as before) is given if there is still fever within 24 hours after the first dose and the interval between two medications ≥ 12 hours.Intravenous infusion, The maximum of cumulative number is two, and the maximum single dose does not exceed 800mg.
  Interventions: Drug: Favipiravir Combined With Tocilizumab
- Favipiravir group (Active Comparator): On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 7 days.
  Interventions: Drug: Favipiravir
- Tocilizumab group (Active Comparator): The first dose is 4 ~ 8mg/kg and the recommended dose is 400mg. For fever patients, an additional application (the same dose as before) is given if there is still fever within 24 hours after the first dose and the interval between two medications ≥ 12 hours.Intravenous infusion, The maximum of cumulative number is two, and the maximum single dose does not exceed 800mg.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Favipiravir Combined With Tocilizumab — Favipiravir: On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 7 days.
  Tocilizumab:The first dose is 4 ~ 8mg/kg and the recommended dose is 400mg. For fever patients, an additional application (the same dose as before) is given if there is still fever within 24 hours after the first dose and the interval between two medications ≥ 12 hours.Intravenous infusion, The maximum of cumulative number is two, and the maximum single dose does not exceed 800mg.
  Arms: Favipiravir Combined With Tocilizumab group
Drug: Favipiravir — On the 1st day, 1600mg each time, twice a day; from the 2nd to the 7th day, 600mg each time, twice a day. Oral administration, the maximum number of days taken is not more than 7 days.
  Arms: Favipiravir group
Drug: Tocilizumab — The first dose is 4 ~ 8mg/kg and the recommended dose is 400mg. For fever patients, an additional application (the same dose as before) is given if there is still fever within 24 hours after the first dose and the interval between two medications ≥ 12 hours.Intravenous infusion, The maximum of cumulative number is two, and the maximum single dose does not exceed 800mg.
  Arms: Tocilizumab group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of favipiravir combined with tocilizumab in the treatment of corona virus disease 2019.

DETAILED DESCRIPTION:
In clinical institutions that enroll patients with corona virus disease 2019, three arms, multi-center, randomized and controlled methods are adopted. Patients are divided into three groups, favipiravir combined with tocilizumab group, favipiravir group and tocilizumab group. 150 patients are expected to be enrolled and the cases are allocated according to the ratio of 3( favipiravir combined with tocilizumab group): 1(favipiravir group): 1(tocilizumab group).

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with Corona Virus Disease 2019
2. Increased interleukin-6
3. Sign the informed consent
4. Subjects who can take medicine orally
5. Agree to collect clinical samples
6. Female subjects of childbearing age are not pregnant and agree to take effective contraception within 7 days of the last oral medication to ensure that they are not pregnant within 3-6 months
7. Male patients agree to effective contraception within 7 days of last oral medication.

Exclusion Criteria:

1. Cases of severe vomiting that make it difficult to take the drug orally
2. Allergic to Favipiravir or tocilizumab
3. Pregnant and lactating women
4. Subjects received specific antiviral drugs such as lopinavir / ritonavir, ribavirin, arbidol, chloroquine phosphate, hydroxychloroquine, and monoclonal antibodies within one week before admission.
5. Cases of respiratory failure and requiring mechanical ventilation
6. Cases of shock
7. Combined organ failure requires ICU monitoring and treatment
8. Predicted clinically that there is no hope of survival, or cases of deep coma that do not respond to supportive treatment measures within three hours of admission
9. Alanine aminotransferase / Aspartate aminotransferase> 5 times of upper limit of normal
10. Neutrophils <0.5 × 10^9 / L, platelets less than 50 × 10^9 / L
11. Clear diagnosis of rheumatoid immunity, malignant tumors and other related diseases
12. Long-term oral anti-rejection drugs or immunomodulatory drugs
13. Allergic reactions to tocilizumab or any excipients
14. Patients with active hepatitis, tuberculosis, and definite bacterial and fungal infections
15. Organ transplant patients
16. Patients with mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-08 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 3 months
  Definition of clinical cure: The viral load of the respiratory specimen was negative for two consecutive times (the interval between the two tests was greater than or equal to one day), the lung image improved, and the body temperature returned to normal for more than 3 days, and the clinical manifestation improved.

SECONDARY OUTCOMES:
Viral nucleic acid test negative conversion rate and days from positive to negative | 14 days after taking medicine
Duration of fever | 14 days after taking medicine
Lung imaging improvement time | 14 days after taking medicine
Mortality rate because of Corona Virus Disease 2019 | 3 months
Rate of non-invasive or invasive mechanical ventilation when respiratory failure occurs | 3 months
Mean in-hospital time | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (6):
- China (6):
  - Guiqiang Wang, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Ezhou Central Hospital, Wuhan, Hubei
  - Huoshenshan Hospital of Wuhan, Wuhan, Hubei
  - Jinyintan Hospital of Wuhan, Wuhan, Hubei
  - Wuhan Pulmonary Hospital, Wuhan, Hubei